CLINICAL TRIAL: NCT02610088
Title: Effect of Dapagliflozin, a Sodium Glucose Co-transporter 2 Inhibitor, on Vascular Functions in Patients With Type 2 Diabetes Compared to Gliclazide
Brief Title: Effect of Dapagliflozin on Vascular Functions in Patients With Type 2 Diabetes Compared to Gliclazide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B-1507/307-006
Record Dates: First submitted 2015-11-15; First posted 2015-11-20 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Diabetes
Keywords: Diabetes; Atherosclerosis; Cardiovascular disease; Endothelial dysfunction; Vascular function; Dapagliflozin; Gliclazide
MeSH Terms: conditions — Diabetes Mellitus; Atherosclerosis; Cardiovascular Diseases | interventions — dapagliflozin; Gliclazide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dapagliflozin (Active Comparator): Dapagliflozin will be started in patient with type 2 diabetes mellitus
  Interventions: Drug: Dapagliflozin
- Gliclazide (Active Comparator): Gliclazide will be started in patient with type 2 diabetes mellitus
  Interventions: Drug: Gliclazide

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10 mg, orally once daily at any time of day with or without food. If HbA1c does not decrease by > 0.4% at 12 week, rescue therapy (sitagliptin 100 mg) can be added at investigator's discretion.
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Gliclazide — Gliclazide MR 30 mg, orally once daily at any time of day with or without food. If HbA1c does not decrease by > 0.4% at 12 week, rescue therapy (gliclazide MR 30 mg) can be added at investigator's discretion.
  Other Names: Diamicron MR
  Arms: Gliclazide

SUMMARY:
The investigators set up a clinical trial to compare effect of dapagliflozin, a sodium glucose co-transporter 2 inhibitor, with gliclazide on vascular function in patients with type 2 diabetes

DETAILED DESCRIPTION:
Obesity, and especially visceral/abdominal adiposity, is associated with diabetes and increased cardiovascular risk. In previous randomized, double-blind, placebo-controlled study, dapagliflozin reduced total body weight, predominantly by reducing fat mass, visceral adipose tissue and sc adipose tissue in type 2 diabetes. This study supported that caloric loss from glycosuria, and not fluid loss, was principally responsible for decrease in total body weight and fat mass. In fact, there have been several reports proving that inhibition of SGLT2 improves β-cell function and reduces body weight and blood pressure. However, effects of SGLT2 inhibitors on lipid profiles have not been decided yet in patients with type 2 diabetes. Furthermore, there are few data to demonstrate the effects of SGLT2 inhibitors on CV risk.

Many systems and pathways are involved in development of atherosclerosis in the arterial wall. Accumulating evidence suggests that endothelial dysfunction plays an important role particularly in the first stage of atherogenesis in patients with diabetes. Approaches designed to improve endothelial function may therefore have additional therapeutic value in the prevention and treatment of atherosclerotic disease. Endothelial dysfunction is related to decreased production and bioavailability of nitric oxide (NO). Endothelial function was measured through several circulating biomarker such as NO, endothelin-1 or non-invasive techniques such as flow-mediated dilation (FMD), skin laser doppler. Among them, FMD is known to as the optimal tool. In addition, several noninvasive techniques including measurement of the ankle-brachial index (ABI), carotid intima-media thickness (IMT) and pulse wave velocity (PWV) have been used for evaluation of atherosclerosis.

If a participant's HbA1c dose not decreas by >0.4% at 12 weeks, rescue therapy can be added at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with HbA1c ≥ 7.5% at screening visit
* Male or female between 40 and 70 years of age
* Patients taking metformin (≥ 1000 mg or maximum tolerated dose) for more than 3 months
* BMI ≥23 kg/m²
* Estimated GFR ≥ 60 ml/min/1.73m²

Exclusion Criteria:

* Patients with acute coronary syndrome within 3 months prior to screening visit
* Pregnant or breast feeding women or reproductive-age women who refuse contraception
* Type 1 diabetes, gestational diabetes, or diabetes with secondary cause
* Chronic hepatitis B or C (except healthy carrier of HBV), liver disease (AST/ALT > 3-fold the upper limit of normal)
* Cancer within 5 years (except squamous cell cancer, cervical cancer, thyroid cancer with appropriate treatment) except thyroid cancer or carcinoma in situ
* Other clinical trial within 30 days
* Alcohol abuse
* Contraindication to SGLT2 inhibitors or sulfonylurea

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Vascular function assessed by Flow-mediated vasodilation (FMD) | 24weeks
  The diameter of the target artery is measured by high-resolution external vascular ultrasound in response to an increase in blood flow (causing shear-stress) during reactive hyperaemia (induced by cuff inflation and then deflation). This leads to endothelium-dependent dilatation; the response is contrasted with that to sublingual nitroglycerin, an endothelium-independent dilator. The artery is scanned and the diameter measured during three conditions; at baseline, during reactive hyperaemia (induced by inflation and then deflation of a sphygmomanometer cuff around the limb, distal to the scanned part of the artery) and finally after administration of sublingual nitroglycerin (which causes endothelium-independent smooth muscle mediated vasodilatation).

SECONDARY OUTCOMES:
Change of blood pressure | 24weeks
Lipid metabolism assessed by triglyceride, low density lipoprotein-cholesterol and high density lipoprotein-cholesterol | 24weeks
Inflammatory markers assessed by hsCRP | 24weeks
Change of body composition assessed by bioelectrical impedance analysis (BIA) methods | 24weeks
Glucose metabolism assessed by glycated hemoglobin and fasting plasma glucose | 24weeks
Microcirculation assessed by laser doppler | 24weeks
Vascular health assessment by pulse wave velocity (PWV) | 24weeks
  PWV, by definition, is the distance traveled (Delta x) by the wave divided by the time (Delta t) for the wave to travel that distance
Vascular health assessment by Ankle-brachial index (ABI) | 24weeks
  The ankle-brachial pressure index (ABPI) or ankle-brachial index (ABI) is the ratio of the blood pressure at the ankle to the blood pressure in the upper arm (brachium).
Carotid intima-media thickness (cIMT) assessed by ultrasound | 24weeks
  Intima-media thickness (IMT), also called intimal medial thickness, is a measurement of the thickness of tunica intima and tunica media, the innermost two layers of the wall of an artery.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea